CLINICAL TRIAL: NCT06611150
Title: A Phase I Study of Concurrent Nab-paclitaxel with Intensity-modulated Radiation Therapy in Patients with Stage III-IVa Nasopharyngeal Carcinoma
Brief Title: Concurrent Nab-paclitaxel with Intensity-modulated Radiation Therapy in Patients with Stage III-IVa Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Fang-Yun Xie, professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2024-076-01
Record Dates: First submitted 2024-09-23; First posted 2024-09-24 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Nasopharyngeal Carcinoma (NPC)
Keywords: nasopharyngeal carcinoma; nab-paclitaxel; concurrent chemotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- nab-paclitaxel arm (Experimental): All patients enrolled in the study will be treated with nab-paclitaxel during radical radiotherapy following induction chemotherapy. The doses are increased progressively from 180 mg/m² to a maximum of 260 mg/m².
  Interventions: Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Nab-paclitaxel — All participants enrolled in the study will be treated with nab-paclitaxel during radical radiotherapy following induction chemotherapy. The doses are increased progressively (180 mg/m², 200 mg/m², 230 mg/m², and 260 mg/m²).

SUMMARY:
The goal of this clinical trial is to determine the maximum tolerated dose and the recommended phase II dose for nab-paclitaxel when administered concurrently with radiotherapy in nasopharyngeal carcinoma. Researchers will observe the toxicity response of patients receiving nab-paclitaxel at 180 mg/m², 200 mg/m², 230 mg/m², and 260 mg/m².

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed nasopharyngeal carcinoma
* III-IVa (AJCC8th)
* age 18-70
* PS score 0-1
* normal functions to tolerate chemotherapy and radiotherapy

Exclusion Criteria:

* The presence of other malignant neoplasms within the preceding five years, with the exception of carcinoma in situ, adequately treated non-melanoma skin cancer and papillary thyroid cancer, is permitted.
* Symptomatic heart failure, unstable angina, myocardial infarction, active infections requiring systemic therapy, psychiatric disorders, or family and social factors

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-08-02 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
The maximum tolerated dose and the recommended phase II dose | From start of radiotherapy to 2 weeks after completion of radiotherapy
  The maximum tolerated dose and the recommended phase II dose for nab-paclitaxel when administered concurrently with radiotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No